CLINICAL TRIAL: NCT00778037
Title: An Open Label, Balanced, Randomized, Two-Treatment, Two-Sequence, Two-Period, Single-Dose, Crossover, Bioavailability Study Comparing Cyclobenzaprine Hydrochloride 10 mg Tablet of Ohm Labs Inc (A Subsidiary of Ranbaxy Pharmaceuticals Inc USA.) With Flexeril® 10 mg Tablet (Containing Cyclobenzaprine Hydrochloride 10 mg) Manufactured by Merck & Co Inc., USA and Distributed by McNeil Consumer & Speciality Pharmaceuticals, in Healthy, Adult, Male, Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Cyclobenzaprine Hydrochloride 10 mg Tablets, USP Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 125_CYCLO_06
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Cyclobenzaprine hydrochloride 10 mg tablet fasting conditions
MeSH Terms: interventions — cyclobenzaprine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cyclobenzaprine hydrochloride 10 mg tablet of ranbaxy
  Interventions: Drug: Cyclobenzaprine hydrochloride 10 mg tablet
- 2 (Active Comparator): Flexeril® 10 mg tablets
  Interventions: Drug: Cyclobenzaprine hydrochloride 10 mg tablet

INTERVENTIONS:
Drug: Cyclobenzaprine hydrochloride 10 mg tablet

SUMMARY:
To compare the single-dose oral bioavailability of Cyclobenzaprine hydrochloride 10 mg tablet of Ohm Labs Inc (A subsidiary of Ranbaxy Pharmaceuticals Inc USA.) with Flexeril® 10 mg tablet (containing Cyclobenzaprine hydrochloride 10 mg) of McNeil Consumer & Specialty Pharmaceuticals, in healthy, adult, male, human subjects under fasting condition.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomized, two-treatment, two-sequence, two-period, single-dose, crossover, bioavailability study comparing Cyclobenzaprine hydrochloride 10 mg tablet of Ohm Labs Inc (A subsidiary of Ranbaxy Pharmaceuticals Inc USA.) with Flexeril® 10 mg tablet (containing Cyclobenzaprine hydrochloride 10 mg) manufactured by Merck & Co Inc., USA and distributed by McNeil Consumer & Speciality Pharmaceuticals, in healthy, adult, male, human subjects under fasting condition.

Following an overnight fast of at least 10 hours, A single oral dose of one Cyclobenzaprine hydrochloride 10 mg tablet was administered with 240 mL of drinking water at ambient temperature during each period of the study under supervision of a trained Study Personnel.

During the course of the study safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical parameters, serology and urine analysis) at baseline. Laboratory parameters of hematology and biochemistry were repeated at the end of the study.

A total of forty (40) subjects were enrolled in the study. Out of which thirty-four (34) subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

* Were in the age range of 18-45 years.
* Were neither overweight nor underweight for his height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

* - Hypersensitivity or allergy to Cyclobenzaprine hydrochloride or related group of drugs.
* Use of MAO Inhibitors in the past 2 weeks / history of Hyperthyroidism.
* History of hypotension, dizziness, syncope or those who had previously experienced a hypotensive response to other medications.
* History of arrhythmia, heart block or congestive heart failure.
* History of urinary disorders especially urinary retention.
* History of seizures, tinnitus, tremors, visual disorders, psychosomatic illness, recurrent palpitations, Jaundice.
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
* Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), epithelial cells (>4/HPF), glucose (positive) or protein (positive).
* Clinically abnormal ECG or Chest X-ray.
* History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or hematological disease, diabetes, glaucoma or increased intra ocular pressure.
* History of any psychiatric illness which might impair the ability to provide written informed consent.
* Regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
* Used any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Participated in any clinical trial within 12 weeks preceding Day 1 of this study.
* Subjects who, through completion of this study, would have donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2006-09 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy CPU, Gurgaon, Haryana, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html